CLINICAL TRIAL: NCT07363005
Title: Effects of a Parent-Child Mandala Painting Intervention During Chemotherapy on Caregiver Burden, Psychological Well-being, and Child Fear and Pain: A Randomized Controlled Trial
Brief Title: Parent-Child Mandala Painting During Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Rıdvan Akdogan, Assist. Prof. (PhD), Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: YYU-MANDALA-ONCO-01
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Childhood Cancers; Pediatric Oncology
Keywords: Mandala painting; Art therapy; Pediatric chemotherapy; Caregiver burden; Child fear; Pain management; Non-pharmacological intervention; Parent-child interaction
MeSH Terms: conditions — Caregiver Burden; Agnosia

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either an intervention group receiving a parent-child mandala painting activity in addition to routine care or a control group receiving routine care alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandala Painting Group (Experimental): Participants in this arm receive a structured parent-child mandala painting intervention in addition to routine nursing care during the chemotherapy process. The intervention is delivered over two weeks, consisting of six sessions, each lasting approximately 30 minutes.
  Interventions: Behavioral: Parent-Child Mandala Painting Intervention
- Control Group (No Intervention): Participants in this arm receive routine nursing care during the chemotherapy process without any additional structured intervention during the study period.

INTERVENTIONS:
Behavioral: Parent-Child Mandala Painting Intervention — This behavioral intervention involves structured parent-child mandala painting sessions conducted during the chemotherapy process. The intervention aims to support children's emotional well-being and fine motor skills while enhancing parent-child interaction. Sessions are delivered over a two-week period, with a total of six sessions, each lasting approximately 30 minutes, and are facilitated by a trained nurse.
  Arms: Mandala Painting Group

SUMMARY:
This randomized controlled trial aims to evaluate the effects of a parent-child mandala painting intervention conducted during the chemotherapy process on caregiver burden, psychological well-being, and child fear and pain levels in pediatric oncology patients.

Childhood cancer and its treatment are highly stressful experiences for both children and their parents. Chemotherapy-related side effects such as pain, fear, and emotional distress may negatively affect children's psychological well-being and treatment adaptation. Parents, as primary caregivers, often experience increased emotional burden, anxiety, and stress during this process.

The intervention consists of a structured parent-child mandala painting activity delivered over a two-week period, with six sessions in total, each lasting 30 minutes. Participants are randomly assigned to either the intervention group, which receives the mandala painting activity in addition to routine care, or the control group, which receives routine nursing care alone.

Outcome measures include child fear and pain levels assessed using validated pediatric scales, as well as caregiver burden and psychological distress measured through standardized questionnaires. Assessments are conducted at baseline and after completion of the two-week intervention period.

This study seeks to contribute evidence on the use of creative, non-pharmacological interventions to support emotional well-being in children undergoing chemotherapy and their caregivers.

DETAILED DESCRIPTION:
This study is designed as a randomized controlled trial to examine the effects of a parent-child mandala painting intervention during the chemotherapy process on caregiver burden, psychological well-being, and child fear and pain levels.

The study population consists of children aged 5-12 years who are receiving chemotherapy treatment in a pediatric hematology-oncology unit and their primary caregivers. Following eligibility screening and informed consent, eligible parent-child dyads are randomly assigned to either the intervention group or the control group using an urn randomization method to ensure equal allocation.

Participants in the intervention group engage in a parent-child mandala painting activity in addition to routine nursing care. The intervention is delivered over a two-week period, consisting of six sessions, each lasting approximately 30 minutes. During each session, children and their parents are provided with mandala coloring sheets and colored markers and are encouraged to paint together in a quiet and supportive hospital environment. The activity aims to promote emotional expression, relaxation, and positive parent-child interaction during chemotherapy.

The control group receives routine nursing care without any additional structured intervention during the same two-week period. After completion of outcome assessments, participants in the control group are also offered the mandala painting activity in accordance with ethical principles.

Primary outcome measures include child fear and pain levels, assessed using the Child Fear Scale and the Wong-Baker Faces Pain Rating Scale. Secondary outcome measures include caregiver burden and psychological distress, measured using the Zarit Caregiver Burden Scale and the Depression Anxiety Stress Scale (DASS-21).

Outcome assessments are conducted at baseline prior to the intervention and at the end of the two-week intervention period. Data are analyzed to compare changes in outcome measures between the intervention and control groups.

This study aims to provide evidence regarding the effectiveness of a non-pharmacological, creative intervention in reducing psychological distress and improving emotional well-being among children undergoing chemotherapy and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 5 and 12 years who are receiving chemotherapy.
* One parent or primary caregiver willing to participate with the child.
* Ability of the child to perform basic fine motor activities such as holding a pencil and coloring.
* Absence of an acute psychiatric diagnosis in the child (e.g., severe anxiety disorder, psychotic disorders).
* Willingness of both the child and the parent to participate in the study.

Exclusion Criteria:

* Children diagnosed with stage III or stage IV cancer.
* Presence of visual perception impairments in the child (e.g., color blindness, severe visual impairment).
* Refusal of the child or parent to participate in the study.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2025-11-22 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Children's Pain Level | Baseline and at the end of the 2-week intervention period
  Change in children's pain level measured using the Wong-Baker Faces Pain Rating Scale (WBFPRS), a validated pediatric pain assessment tool consisting of six facial expressions representing increasing pain intensity. The scale is scored from 0 to 10, where 0 indicates "no pain" and 10 indicates "worst pain imaginable." Higher scores represent greater pain intensity.
Children's Fear Level | Baseline and at the end of the 2-week intervention period
  Change in children's fear level measured using the Children's Fear Scale (CFS), a single-item observational scale designed to assess fear in children. The scale ranges from 0 to 4, where 0 represents "no fear" and 4 represents "extreme fear." Higher scores indicate higher levels of fear.

SECONDARY OUTCOMES:
Caregiver Burden | Baseline and at the end of the 2-week intervention period
  Change in caregiver burden measured using the Zarit Burden Interview (ZBI), a widely used self-report questionnaire assessing the perceived burden of caregivers. The scale consists of 22 items with total scores ranging from 0 to 88, where higher scores indicate greater caregiver burden.
Parental Psychological Distress | Baseline and at the end of the 2-week intervention period
  Change in parental psychological distress measured using the Depression Anxiety Stress Scale-21 (DASS-21), a self-report instrument assessing symptoms of depression, anxiety, and stress. Total scores range from 0 to 63, with higher scores indicating greater psychological distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yuzuncu Yil University Dursun Odabas Medical Center, Van, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the sensitive nature of the study population, which includes pediatric patients undergoing chemotherapy and their caregivers. The data contain personal and psychological assessment information, and sharing IPD could pose risks to participant privacy and confidentiality.